CLINICAL TRIAL: NCT06254924
Title: Qoyangnuptu: QI App Pilot for Assessing Feasibility and Acceptability of a Mobile Health App for Adolescents in a Southwestern Tribal Community
Brief Title: Qoyangnuptu: Qoyangnuptu Intervention (QI) App
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2125143
Record Dates: First submitted 2024-01-29; First posted 2024-02-12 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Wellness 1
Keywords: American Indian / Alaska Native; mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QI App Users (Experimental): Participants will be asked to use the QI App once per day for 5-10 minutes per day for 6 weeks.
  Interventions: Behavioral: QI App Users
- Parents/Guardians of QI App Users (Experimental): Parents/guardians of QI App users will be aware that their child is using the QI App once per day for 5-10 minutes per day for 6 weeks.
  Interventions: Behavioral: Parents/Guardians of QI App Users

INTERVENTIONS:
Behavioral: QI App Users — QI App users will be asked to complete a daily, 2-question mood and stress survey. They will be encouraged to use the QI App to practice mindfulness skills including meditation, drawing, coloring, breathing, and walking. They will be encouraged to use the QI App to help them participate in asynchronous group running activities.
  Arms: QI App Users
Behavioral: Parents/Guardians of QI App Users — Parents/Guardians of QI App users will be informed that their child is using the QI App for a 6-week period.
  Arms: Parents/Guardians of QI App Users

SUMMARY:
The goal of this clinical trial is to learn about the impacts of using a mobile health app, the Qoyangnuptu Intervention App (QI App) a Southwestern Tribal Community. The main questions it aims to answer are:

In American Indian/Alaska Native communities with unique cultural characteristics, how should a youth-focused sociotechnical behavioral health intervention be designed to encourage sustained engagement and positively impact indicators of behavioral health?; How can interactive technical interventions be designed to best support sustained community engagement in a challenged network environment?

Participants will:

* Receive daily guidance and encouragement to use the app from an anonymous, trained peer mentor
* Be able to ask their peer mentors questions in a monitored one-on-one chat in the QI app or in a monitored group chat in the QI app
* Log their mood and stress level on the app once per day
* Practice mindfulness skills as directed in the QI app, including guided breathing, meditation, drawing, coloring, and walking
* Practice Hopi cultural activities like running using the QI app to help track progress towards team mileage goals

DETAILED DESCRIPTION:
Indigenous youth face behavioral health challenges at much higher rates than non-Indigenous youth in the United States. Some of the reasons for these disparities include lack of culturally responsive behavioral health training and coping resources and lack of access to in-person behavioral health resources and interventions. This research seeks to investigate the impact that a mobile phone app that teaches mindfulness and provides opportunities for mindfulness practice might help adolescents from a Southwestern Tribal community increase measures of resilience. The mobile phone app, called the QI App, has been designed with members of the Southwestern Tribal community to ensure cultural appropriateness and responsiveness. It has also been designed with research experts from clinical psychology, serious game design, and computer networking to ensure that it uses evidence-based best practices.

1. Recruitment The investigators will use a multipronged recruitment strategy. Recruitment will be carried out by the study team's Community Research Coordinator.

   Because the QI App was designed with members of the Southwestern Tribal community as consultants, the investigators already have individual contact information for people who have stated they would like to be reached out to when the investigators are ready to recruit for the pilot. The investigators will use a direct email approach with these individuals.

   Through the QI App design process, the study team encountered a number of individuals and organizations who indicated that they would like to share the recruitment posts on their social media when the time came for the pilot. The investigators will prepare a social media post that potential participants can share on their networks.

   The investigators will work with their community research coordinator and their Senior Personnel and project consultants to help them post flyers strategically in the community.

   When working with Indigenous communities, developing trust is paramount. One of the best ways for the investigators to successfully recruit is for individuals who have come to know and trust the study team reach out to others in their community to share information about the study and have them reach out to contact the study team to be formally recruited. Individuals who reach out to the study team via word-of-mouth will be followed up with using the Email Recruitment message.
2. Consent Process

   Once individuals have made contact with the study team via recruitment effort, the investigators will plan to have a Zoom meeting with potential participants or in a reserved community meeting room to review the study details, answer questions, and obtain informed consent. This meeting will also require the participant to download and install the QI App to demonstrate that they can use it on their personal iPhone or Android device.
   * If meeting over Zoom: The investigators will obtain consent through a Zoom oral consent statement. The investigators will email the consent form to participants or send to them via postal mail if they prefer.
   * If meeting in-person: The investigators will reserve a community room where potential participants can meet with the study team's community researcher at a scheduled time to review the research process in a space that allows for confidentiality to be maintained. Participants will physically sign the consent form and be provided with a copy.
3. Research Activities

   * QI App Users. The participants will be asked to complete a short demographic questionnaire and baseline survey. The participants will be asked to use the QI App for a total for 6 weeks. After the participants have completed the 6-week cohort, they will again complete the QI App user questionnaire (which combines all questionnaire measures for Secondary Study Objectives 1-6 in "Project Purpose" Section). They will also be asked to participate in a focus group with semi-structured interview questions where they will explain what they liked and did not like about the QI App and what they would change about the app and user experience. 12 weeks after the completion of the program (12 weeks from when they started using the app), participants will complete the QI App user questionnaire for the third time. Surveys can be distributed either as electronic surveys sent via email OR via physical delivery and pickup by the community research coordinator, whichever the subject prefers. Focus groups will be conducted either as Zoom sessions or in-person in a reserved community room, depending on the collective preference of participants.
   * Parents of QI App Users. The participants will be asked to complete a short demographic questionnaire and baseline survey.. After the participant's child has completed the 6-week cohort, they will again complete the Parents of QI App user survey (which combines all questionnaire measures for Secondary Study Objectives 7-8 in "Project Purpose" Section). They will also be asked to participate in a focus group with semi-structured interview questions where they will explain what they liked and did not like about the QI App and what they would change about the app and user experience.12 weeks after the completion of the program (12 weeks from when they started using the app), participants will complete the QI App user questionnaire for the third time. Surveys can be distributed either as electronic surveys sent via email OR via physical delivery and pickup by the community research coordinator, whichever the subject prefers. Focus groups will be conducted either as Zoom sessions or in-person in a reserved community room, depending on the collective preference of participants.

ELIGIBILITY:
Inclusion Criteria:

* 14-25 years old
* Belongs to Southwestern Tribal community
* Has a smartphone capable of running the QI App
* Is able to access the Internet with smartphone at least once per day

Exclusion Criteria:

* Younger than 14 or older than 25
* Does not belong to Southwestern Tribal Community
* Does not have a smartphone capable of running the QI App
* Is not able to access the Internet with smartphone at least once per day

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
To measure the acceptability of the QI App. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  Through qualitative interviews, the investigators will determine the acceptability of the QI App. 12 participants will be interviewed after they have used the app for 6 weeks.

SECONDARY OUTCOMES:
Impact of app usage on attitudes towards seeking professional mental health assistance. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  Measured by the Attitudes Towards Seeking Professional Psychological Help - Short Form Scale before participating as a Peer Mentor, 6 weeks into participating as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Attitudes Towards Seeking Professional Psychological Help is a 10-item measure used to assess attitudes towards seeking professional psychological help on a 4-point Likert scale, ranging from 0 to 3. Higher total score indicates more positive attitudes towards seeking seeking professional psychological help and is associated with lower levels of stigma against mental illness.
Impact of app usage on measures of depression. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  Patient Health Questionnaire-9 before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Patient Health Questionnaire-9 is a 9-item measure used to assess frequency that a participant experiences depressive symptoms. Each item is score on a 4-point scale from 0 ("not at all") to 3 ("every day"). Higher total scores indicate more frequent experience of depressive symptoms.
Impact of app usage on measures of stress. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  Perceived Stress Scale 4 before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Perceived Stress Scale 4 measures participant perceptions of their thoughts and feelings over the past month on 4 items. Each item is scored on a 5-point scale from from 0 ("Never") to 4 ("Very Often"). Higher scores indicate higher levels of stress.
Impact of app usage on measures of mindfulness. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  State Mindfulness Scale Physical Activity before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The State Mindfulness Physical Activity scale is a 12 item measure with six items assessing state mindfulness of the mind (i.e., thoughts and emotions) and six items assessing state mindfulness of the body (i.e., movement, body sensations, muscle engagement). The response scale is 0 - 4, with anchors of Not at all (0) and Very much (4). Initial evidence supports a bi-factor structure of the measure in which both a general state mindfulness factor and two specific factors (mind and body) are supported. The bi-factor structure supports the use of using a single score to capture overall state mindfulness, but also the use of two scores capture mindfulness of the mind and mindfulness of the body.
Impact of app usage on measures of quiet ego. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  Quiet Ego Scale before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Quiet Ego Scale is a 14 item measure that assesses detached awareness, inclusive identity, perspective taking, and growth. Each item is assessed on a 5-point Likert scale from 1 ("strongly disagree") to 5 ("strongly agree"). A higher score indicates a stronger quiet ego.
Impact of app usage on measures of social connectedness. | Baseline, 6 weeks after starting the app, 12 weeks after starting the app
  University of California Los Angeles Loneliness Scale 3 before participating as a Peer Mentor, 6 weeks into participation as a Peer Mentor, and 12 weeks after starting as a peer mentor.
  The Loneliness Scale 3 comprises 3 questions that measure 3 dimensions of loneliness: relational connectedness, social connectedness, and self-perceived isolation. Each item is measured on a 3-point scale from 1 ("Hardly Ever") to 3 ("Often"). Higher scores indicate greater perceptions of loneliness.
Impact of child's usage of QI App on parent/guardian attitudes towards seeking professional mental health assistance. | Baseline, 6 weeks after starting the app, 12 weeks after child starts using the app
  Measured by the Attitudes Towards Seeking Professional Psychological Help - Short Form Scale before participant's child starts using the QI App, 6 weeks after participant's child starts using the QI App, and 12 weeks after the participant's child starts using the QI App.
  The Attitudes Towards Seeking Professional Psychological Help is a 10-item measure used to assess attitudes towards seeking professional psychological help on a 4-point Likert scale, ranging from 0 to 3. Higher total score indicates more positive attitudes towards seeking seeking professional psychological help and is associated with lower levels of stigma against mental illness.
Impact of child's usage of QI App on parent/guardian perceptions of their child's behavior and emotions. | Baseline, 6 weeks after starting the app, 12 weeks after participant's child starts using the app.
  Measured by the Child Behavior Checklist.
  The Child Behavior Checklist 6-18 has parents assess both child adaptive behaviors and problem behaviors. There are 112 items that assess problem behaviors and 20 items that assess adaptive behavior. Response format for problem behaviors is from 0 ("not true") to 2 ("very true"). A Total Competence and Total Behavior Problems score are also provided. Higher scores of Total Competence indicate that the child being evaluated has a greater number of adaptive behaviors. Higher scores of Total Behavior Problems indicate greater incidence of problem behaviors observed associated with the child being evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Vigil-Hayes, PhD, Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Given the small population from which we will be recruiting, releasing IPD could inadvertently compromise confidentiality.

REFERENCES:
- [Background] Vigil-Hayes M, Collier AF, Hagemann S, Castillo G, Mikkelson K, Dingman J, Munoz A, Luther J, McLaughlin A. Integrating Cultural Relevance into a Behavioral mHealth Intervention for Native American Youth. Proc ACM Hum Comput Interact. 2021 Apr;5(CSCW1):165. doi: 10.1145/3449239. PMID 34676359
- [Background] Vigil-Hayes M, Futterman Collier A, Castillo G, Blackhorse D, Awbery N, Abrahim JP. Designing a Mobile Game That Develops Emotional Resiliency in Indian Country. Ext Abstr Hum Factors Computing Syst. 2019 May;2019:LBW2122. doi: 10.1145/3290607.3312790. PMID 32455346
- [Background] Picco L, Abdin E, Chong SA, Pang S, Shafie S, Chua BY, Vaingankar JA, Ong LP, Tay J, Subramaniam M. Attitudes Toward Seeking Professional Psychological Help: Factor Structure and Socio-Demographic Predictors. Front Psychol. 2016 Apr 25;7:547. doi: 10.3389/fpsyg.2016.00547. eCollection 2016. PMID 27199794
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Cox AE, Ullrich-French S, Howe HS, Cole AN. A pilot yoga physical education curriculum to promote positive body image. Body Image. 2017 Dec;23:1-8. doi: 10.1016/j.bodyim.2017.07.007. Epub 2017 Aug 14. PMID 28818786
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Achenbach TM, Ruffle TM. The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatr Rev. 2000 Aug;21(8):265-71. doi: 10.1542/pir.21-8-265. No abstract available. PMID 10922023